CLINICAL TRIAL: NCT07025382
Title: Relative Effect of Home-based Telerehabilitation Compared to Center-based Pulmonary Rehabilitation for Patients With Chronic Obstructive Pulmonary Disease: A Multicenter Randomized Controlled Non-inferiority Study
Brief Title: Telerehabilitation Versus Centre-based Pulmonary Rehabilitaztion for Patients With Chronic Obstructive Pulmonary Disease
Acronym: TELEREHA-COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ADIR Association (Other)
Collaborators: Région Normandie (Other Government); Département de la Seine Maritime (Unknown); European Union (Other); Centre Hospitalier des Pays de Morlaix (Other); Hopital La Musse (Other); Groupe Hospitalier du Havre (Other); Groupe Havrais d'Aide aux Handicapés Respiratoires (Unknown); Union des Kinésithérapeutes et des Rééducateurs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TELEREHA-COPD
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Telerehabilitation; Pulmonary rehabilitation; Center-based exercise training; Home-based exercise training; Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized non-inferiority trial with concealed allocation, a blinded assessor, and an intention-to-treat analysis.
Who Masked: Outcomes Assessor
Masking Description: Statistician wil be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based pulmonary rehabilitation (Experimental): 24 home-based pulmonary rehabilitation sessions
  Interventions: Other: Home-based pulmonary rehabilitation
- Center-based pulmonary rehabilitation (Active Comparator): 24 center-based pulmonary rehabilitation sessions
  Interventions: Other: Center-based pulmonary rehabilitation

INTERVENTIONS:
Other: Home-based pulmonary rehabilitation — An eight-week (three sessions per week) telerehabilitation home-based program, including:
  Twenty-four PR sessions (approximately 1 hour 45 minutes each), including a 15-minute warm-up period, endurance training on a cycle ergometer, muscle strengthening exercises, balance exercises, as well as therapeutic patient education sessions tailored to the patient's needs based on the initial assessment. Training is adjusted according to patient tolerance and healthcare professional recommendations. Participants will receive a cycle ergometer, pulse oximeter, activity tracker, and a tablet application (TELEREHAPP) for guidance throughout the program, remote monitoring, and communication. Home-based sessions include:
  * Endurance training on the cycle ergometer (15 to 45 minutes per session).
  * Strength training and balance exercises (30 minutes per session).
  * Physical activity coaching, including a daily step goal.
  Arms: Home-based pulmonary rehabilitation
Other: Center-based pulmonary rehabilitation — An eight-week (three sessions per week) center-based pulmonary rehabilitation program, including:
  Twenty-four center-based PR sessions (approximately 1 hour 45 minutes each), including a 15-minute warm-up period, endurance training on a cycle ergometer, muscle strengthening exercises, balance exercises, as well as therapeutic patient education sessions tailored to the patient's needs based on the initial assessment. Training is adjusted according to patient tolerance and healthcare professional recommendations.
  Arms: Center-based pulmonary rehabilitation

SUMMARY:
Background and study aims:

Chronic obstructive pulmonary disease is a leading cause of mortality worldwide. Pulmonary rehabilitation is recommended for patients to improve dyspnea, exercise capacity, and quality of life. Paradoxically, as few as 5 to 10% of eligible patients undergo pulmonary rehabilitation due to barriers such as transportation difficulties and limited availability of pulmonary rehabilitation centers. Home-based pulmonary rehabilitation using advanced telehealth technologies (telerehabilitation) may offer a solution to improve access.

This study aims to compare the relative effectiveness of a home-based telerehabilitation program with center-based program. The primary objective is to assess changes in exercise endurance capacity, measured by endurance time, before and after participation of the rehabilitation program.

Who can participate?

Adults between 45 and 80 years old who are referred for pulmonary rehabilitation and have a confirmed diagnosis of chronic obstrucitve pulmonary disease (GOLD stage II to IV) at any of the participating centers are eligible to participate, whether or not they use oxygen during exercise. Participants must live at home with another adult who is present during exercise sessions. They must not have experienced any exacerbation in the month prior to study inclusion, nor have participated in a pulmonary rehabilitation program within the past year. Participants must not have any scheduled surgery within the next four months, including surgery for lung cancer resection. They must not have active cancer, and must not present any contraindication to exercise or any condition that would limit their ability to use the telerehabilitation system.

Eligible participants must be beneficiaries of a social security system and must have read and understood the information letter and signed the informed consent form.

What does the study involve?

This is a multi-center, randomized controlled trial with two groups:

Center-based rehabilitation group: Participants will attend 24 sessions over eight weeks (three sessions per week) at the center. The program includes an initial session of therapeutic education and exercise training, followed by 24 rehabilitation sessions, and a final assessment with educational reinforcement.

Home-based rehabilitation group: Participants will have 24 sessions at home over the same period (eight weeks). The program includes an initial in-center assessment session, followed by 24 rehabilitation sessions and a final in-center session for assessment. They will be provided with equipment such as a cycle ergometer, pulse oximeter, physical activity tracker, and a tablet application (TELEREHAPP) to guide and monitor their home-based exercises. Regular phone contact with healthcare professionals will be maintained for support.

All participants will undergo assessments before and after the program, including a constant work rate endurance test on a cycle ergometer to measure exercise endurance capacity.

What are the possible benefits and risks of participating?

Participants may experience improved physical fitness, which could lead to better dyspnea management and better quality of life. Risks may include muscle soreness, fatigue, or injury related to exercise, independently of group allocation. All exercise sessions will be supervised or monitored to minimize these risks. Participants will receive instructions on how to perform exercises safely and will be encouraged to report any adverse effects promptly.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease is a disabling respiratory condition and a leading cause of mortality worldwide. Suggested treatments are mainly symptomatic and aim to stabilize the progression of the disease. However, a major consequence of COPD is reduced exercise tolerance, which can lead patients to avoid physical activity, further inducing progressive muscle deconditioning and disabling dyspnea.

Pulmonary rehabilitation is recommended by leading international respiratory societies as a core component of the treatment for people with chronic obstructive pulmonary disease. The effectiveness of pulmonary rehabilitation is well established, with numerous studies showing that it improves dyspnea, exercise capacity, quality of life, as well as it reduces mortality and hospital length of stay following exacerbations.

Paradoxically, as few as 5 to 10% of eligible patients undergo pulmonary rehabilitation. Some known barriers to uptake include transportation difficulties and the limited availability of PR centers.

Telerehabilitation may offer an alternative to traditional center-based programs. Results from studies evaluating the clinical benefits of telerehabilitation suggest that it is non-inferior to traditional center-based pulmonary rehabilitation. However, the clinical outcomes reported for the control groups (center-based programs) in these studies were lower than those reported in the reference meta-analysis by McCarthy et al. (2015), which established the benefits of pulmonary rehabilitation, making interpretation of the results difficult. For these reasons, it remains important to continue investigating and comparing these two different modalities.

This study primarily aims to evaluate the relative effect of a 24-session home-based telerehabilitation program compared to a center-based program in patients with chronic obstructive pulmonary disease. The primary outcome is the change in endurance exercise capacity. Secondary outcomes include changes in maximal exercise capacity, functional capacity, quadriceps maximal isometric strength, functional dyspnea, physical activity, sleep quality, self-efficacy, patient autonomy, quality of life, psychological and health status, and cognitive function. Additional outcomes include adherence, environmental impact, a health economic analysis, and a 1-year follow-up to assess hospitalizations, exacerbations, and mortality as well as others outcomes.

Study design :

This is a prospective, multicenter, randomized controlled non-inferiority trial with concealed allocation and a single-blind design (blinded evaluator). Participants will be randomly assigned to one of two groups:

Center-based pulmonary rehabilitation group (24 sessions in total over 8 weeks) : participants will attend 26 center-based visits, over eight weeks, comprising:

* One initiation center-based visit(approximately 3 hours), including an initial assessment by a blinded assessor, self management diagnostic, endurance training on a cycle ergometer, strength training, balance exercises and a leaflet containing educational information and exercise recommendations to guide the patient toward full autonomy.
* Twenty-four center-based PR sessions (approximately 1 hour 45 minutes each), including a 15-minute warm-up period, endurance training on a cycle ergometer, muscle strengthening exercises, balance exercises, as well as therapeutic patient education sessions tailored to the patient's needs based on the initial assessment. Training is adjusted according to patient tolerance and healthcare professional recommendations as follow :
* Endurance training on the cycle ergometer (15 to 45 minutes per session).
* Strength training and balance exercises (30 minutes per session).
* Physical activity coaching.
* Self management at the center (before or after exercise session).
* One final center-based visit (approximately 3 hours), including a final assessment by a blinded assessor, a program review, and educational reinforcement.

Home based telerehabilitation group (24 sessions in total over 8 weeks) : participants will attend 2 visits at the center and perform 24 sessions at home, over eight weeks, comprising:

* One initiation center-based visit (approximately 3 hours), including an initial assessment by a blinded assessor, self management diagnostic, endurance training on a cycle ergometer, strength training, balance exercises and a leaflet containing educational information and exercise recommendations to guide the patient toward full autonomy as well as patient education on how to use the telerehabilition system.
* Twenty-four PR sessions (approximately 1 hour 45 minutes each), including a 15-minute warm-up period, endurance training on a cycle ergometer, muscle strengthening exercises, balance exercises, as well as therapeutic patient education sessions tailored to the patient's needs based on the initial assessment. Training is adjusted according to patient tolerance and healthcare professional recommendations. Participants will receive a cycle ergometer, pulse oximeter, activity tracker, and a tablet application (TELEREHAPP) for guidance throughout the program, remote monitoring, and communication. Home-based sessions include:
* Endurance training on the cycle ergometer (15 to 45 minutes per session).
* Strength training and balance exercises (30 minutes per session).
* Physical activity coaching, including a daily step goal.
* Regular remote monitoring and support via the tablet application, with weekly check-ins from healthcare professionals.
* Self management through videoconferencing.
* One final center-based session (approximately 3 hours), including a final assessment by a blinded assessor, a program review, and educational reinforcement.

Sample size calculation for non-inferiority study:

Assuming a mean difference of 0 seconds between the two groups in the constant work rate endurance test, a non-inferiority margin of 105 seconds, a conservative standard deviation of 150 seconds, an alpha risk of 0.05, and a beta risk of 0.05, a total of 45 patients per group will be needed, totaling 90 patients.

Statistical analysis:

Categorical data will be presented as counts (percentages). Continuous descriptive data will be expressed as means (standard deviation) or medians (interquartile range), depending on their distribution. The normality of distributions will be assessed using the Kolmogorov-Smirnov test.

The analysis will be performed on an intention-to-treat basis using the last observation carried forward method. A per-protocol sensitivity analysis will also be conducted.

The relative effect of the interventions on the primary outcome and other outcomes with repeated measures will be analyzed using a mixed linear model with group (telerehabilitation or center-based rehabilitation), time of measurement (start and end of the program, 1-year follow-up), and their interaction as fixed effects factors, and participant as a random effect factor. Based on available data from the literature, analyses will be adjusted for age, use of long-term oxygen therapy, baseline 6-minute walk distance (except for analyses already including the 6MWD), functional dyspnea (except for analyses already including dyspnea), Forced Expiratory Volume in 1 Second, number of hospitalizations in the past 12 months, anxiety and depression scores (except for analyses already including these outcomes), as well as health status (except for the analysis already including this outcome).

The relative effect of the interventions on outcomes assessed only at the end of the program (e.g. environmental analysis) will be analyzed using a linear mixed model with group (telerehabilitation or center-based rehabilitation) as a fixed effect factor and participant as a random effect factor. The analysis concerning VO₂ peak will be adjusted for the same covariates as the primary outcome.

The difference in effect between groups will be expressed as a mean difference (95% CI) and interpreted according to the minimal clinically important difference specific to each outcome measure, when available in the literature.

The relative effect of the interventions on health events (exacerbations, hospitalizations, death) and program adherence will be assessed using the relative risk at 1 year (95% CI) and adjusted using the same covariates as for the primary outcome analysis. The hazard ratio for time to first exacerbation or death will also be estimated.

Health economic analysis:

Differences in costs and outcomes will be estimated using the seemingly unrelated regression method. These differences will be adjusted using the same covariates as those used in the clinical analyses of the primary outcome, in addition to the randomization arm and baseline utility score for quality-adjusted life years.

A non-parametric bootstrap will be used to represent uncertainty related to estimates for cost-effectiveness.

Analyses will be performed using GraphPad 8 and R software.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 80 years
* Confirmed diagnosis of chronic obstructive pulmonary disease, GOLD stage II to IV
* Stable condition (no exacerbation in the last month prior to participation)
* Referred to a pulmonary rehabilitation program
* With or without oxygen during exercise
* No pulmonary rehabilitation program in the last 12 months prior to participation
* Living at home with another adult present during exercise sessions
* Affiliated with a health insurance system
* Able to read and understand the information letter and sign the consent form

Non-inclusion criteria:

* Referred to pulmonary rehabilitation before lung cancer surgery
* Referred to pulmonary rehabilitation before lung volume reduction surgery scheduled within the next four months
* Visual, cognitive, or auditory impairments incompatible with participation in a tele-pulmonary rehabilitation program
* Orthopedic, neurological, cardiovascular, or neuromuscular conditions limiting exercise training on a cycle ergometer
* Active cancer
* Unable to provide informed consent
* Under legal guardianship or curatorship
* Pregnant or breastfeeding women

Exclusion Criterion:

* Withdrawal of consent

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Endurance time | 2 months
  Endurance time will be assessed during a constant work rate endurance test (75% of peak power output) on a cycle ergometer before and after the prehabilitation program and after 1 year of the enrollement date. The pre-specified minimal clinically important difference is set at 105 seconds.

SECONDARY OUTCOMES:
Endurance time | One year
  Endurance time will be assessed during a constant work rate endurance test (75% of peak power output) on a cycle ergometer before and after the prehabilitation program and after 1 year of the enrollement date. The pre-specified minimal clinically important difference is set at 105 seconds.
Peak oxygen uptake | 2 months
  Peak oxygen uptake will be assessed during an incremental cardiopulmonary exercise testing on a cycle ergometer before and after the rehabilitation program.
Peak power output | 2 months
  Peak power output will be assessed during an incremental cardiopulmonary exercise testing on a cycle ergometer before and after the rehabilitation program.
Functional capacity | 2 months
  Functional capacity will be assessed using the six-minute-walk test before and after the rehabilitation program and after 1 year of the enrollement date. The pre-specified minimal clinically important difference is set at 25 meters.
Functional capacity | One year
  Functional capacity will be assessed using the six-minute-walk test before and after the rehabilitation program and after 1 year of the enrollement date. The pre-specified minimal clinically important difference is set at 25 meters.
Quadriceps muscle isometric strength | 2 months
  Maximum voluntary quadriceps muscle isometric strength will be assessed by dynamometry before and after the rehabilitation program and after 1 year of the enrollement date. The pre-specified minimal clinically important difference is set at 7.5 Nm.
Quadriceps muscle isometric strength | One year
  Maximum voluntary quadriceps muscle isometric strength will be assessed by dynamometry before and after the rehabilitation program and after 1 year of the enrollement date. The pre-specified minimal clinically important difference is set at 7.5 Nm.
Quality of life - Saint George's Respiratory Questionnaire | 2 months
  Quality of life will be assessed using the Saint George's Respiratory Questionnaire. This self-administered questionnaire ranges from 0 to 100, with higher values indicating greater impairment in health-related quality of life. The established minimal clinically important difference for this questionnaire has been established at -4 points.
Quality of life - Saint George's Respiratory Questionnaire | One year
  Quality of life will be assessed using the Saint George's Respiratory Questionnaire. This self-administered questionnaire ranges from 0 to 100, with higher values indicating greater impairment in health-related quality of life. The established minimal clinically important difference for this questionnaire has been established at -4 points.
Quality of life - Euro-Qol five-dimension five-level questionnaire | 2 months
  Quality of life will be assessed using the Euro-Qol five-dimension five-level (EQ-5D-5L) before and after the rehabilitation program and after 1 year of the enrollement date. The EQ-5D-5L consists of five dimensions, each rated on five levels of severity. Responses are converted into a single utility index score, ranging from less than 0 (representing health states worse than death) to 1 (perfect health), with higher scores indicating better health-related quality of life.
  The EQ visual analogue scale (EQ-VAS), ranging from 0 (worst imaginable health) to 100 (best imaginable health), will also be recorded.
Quality of life - Euro-Qol five-dimension five-level questionnaire | One year
  Quality of life will be assessed using the Euro-Qol five-dimension five-level (EQ-5D-5L) before and after the rehabilitation program and after 1 year of the enrollement date. The EQ-5D-5L consists of five dimensions, each rated on five levels of severity. Responses are converted into a single utility index score, ranging from less than 0 (representing health states worse than death) to 1 (perfect health), with higher scores indicating better health-related quality of life.
  The EQ visual analogue scale (EQ-VAS), ranging from 0 (worst imaginable health) to 100 (best imaginable health), will also be recorded.
Functional dyspnea | 2 months
  Functional dyspnea will be assessed using the modified medical research council (mMRC) scale before and after the rehabilitation program and after 1 year of the enrollement date. The mMRC score ranges from 0 to 4, with lower scores indicating less severe functional dyspnea. The pre-specified minimal clinically important difference is set at -1 point.
Functional dyspnea | One year
  Functional dyspnea will be assessed using the modified medical research council (mMRC) scale before and after the rehabilitation program and after 1 year of the enrollement date. The mMRC score ranges from 0 to 4, with lower scores indicating less severe functional dyspnea. The pre-specified minimal clinically important difference is set at -1 point.
Intensity of dyspnea during exercise | 2 months
  The intensity of dyspnea during constant workload exerice test will be assessed using the 10-Borg scale every 30 second during the test. The intensity of dyspnea will be evaluated using the Borg scale, which ranges from 0 to 10. This scale allows for values between 0 (absence of breathlessness) and 10 (maximal breathlessness). Patients will be asked, "What is the intensity of your breathlessness?" The minimal clinically important difference for this outcome is 1 point.
Intensity of dyspnea during exercise | One year
  The intensity of dyspnea during constant workload exerice test will be assessed using the 10-Borg scale every 30 second during the test. The intensity of dyspnea will be evaluated using the Borg scale, which ranges from 0 to 10. This scale allows for values between 0 (absence of breathlessness) and 10 (maximal breathlessness). Patients will be asked, "What is the intensity of your breathlessness?" The minimal clinically important difference for this outcome is 1 point.
Intensity of lower limb fatigue during exercise | 2 months
  The intensity of lower limb fatigue during constant workload exerice test will be assessed using the 10-Borg scale every 30 second during the test. The intensity of lower limb fatigue will be evaluated using the Borg scale, which ranges from 0 to 10. This scale allows for values between 0 (absence of breathlessness) and 10 (maximal breathlessness). Patients will be asked, "What is the intensity of the fatigue in your legs?" The minimal clinically important difference for this outcome is 1 point.
Intensity of lower limb fatigue during exercise | One year
  The intensity of lower limb fatigue during constant workload exerice test will be assessed using the 10-Borg scale every 30 second during the test. The intensity of lower limb fatigue will be evaluated using the Borg scale, which ranges from 0 to 10. This scale allows for values between 0 (absence of breathlessness) and 10 (maximal breathlessness). Patients will be asked, "What is the intensity of the fatigue in your legs?" The minimal clinically important difference for this outcome is 1 point.
Sensory dimension of dyspnea following exercise | 2 months
  he sensory dimension of dyspnea will be assessed using French version of the Multidimensional Dyspnea Profile questionnaire, taking into account the last 30 seconds of effort during the constant workload exercise test to complete the questionnaire. This self-administered questionnaire can yield scores ranging from 0 to 10, with higher scores indicating a greater sensory dimension of dyspnea. The established minimal clinically important difference for this outcome is 2 points.
Sensory dimension of dyspnea following exercise | One year
  he sensory dimension of dyspnea will be assessed using French version of the Multidimensional Dyspnea Profile questionnaire, taking into account the last 30 seconds of effort during the constant workload exercise test to complete the questionnaire. This self-administered questionnaire can yield scores ranging from 0 to 10, with higher scores indicating a greater sensory dimension of dyspnea. The established minimal clinically important difference for this outcome is 2 points.
Affective dimension of dyspnea following exercise | 2 months
  The affective dimension of dyspnea will be assessed using the french version of the Multidimensional Dyspnea Profile questionnaire, considering the last 30 seconds of effort during the constant workload exercise test to complete the questionnaire. This self-administered questionnaire can yield scores ranging from 0 to 10, with higher scores indicating a significant affective dimension of dyspnea. The established minimal clinically important difference for this outcome is 3 points.
Affective dimension of dyspnea following exercise | One year
  The affective dimension of dyspnea will be assessed using the french version of the Multidimensional Dyspnea Profile questionnaire, considering the last 30 seconds of effort during the constant workload exercise test to complete the questionnaire. This self-administered questionnaire can yield scores ranging from 0 to 10, with higher scores indicating a significant affective dimension of dyspnea. The established minimal clinically important difference for this outcome is 3 points.
Health status | 2 months
  Health status will be assessed using the Chronic obstructive pulmonary disease Assessment Test (CAT) before and after the rehabilitation program and after 1 year of the enrollement date. The score ranges from 0 to 40, with higher values indicating greater impairment of health status. The established minimal clinically important difference for this questionnaire is -2.5 points.
Health status | One year
  Health status will be assessed using the Chronic obstructive pulmonary disease Assessment Test (CAT) before and after the rehabilitation program and after 1 year of the enrollement date. The score ranges from 0 to 40, with higher values indicating greater impairment of health status. The established minimal clinically important difference for this questionnaire is -2.5 points.
Symptoms of anxiety | 2 months
  Symptoms of anxiety will be assessed using the Hospital Anxiety and Depression questionnaire, anxiety subscore, before and after the rehabilitation program and after 1 year of the enrollement date. The score ranges from 0 (best) to 21 (worst). The pre-specified minimal clinically important difference is set at -1.5 point.
Symptoms of anxiety | One year
  Symptoms of anxiety will be assessed using the Hospital Anxiety and Depression questionnaire, anxiety subscore, before and after the rehabilitation program and after 1 year of the enrollement date. The score ranges from 0 (best) to 21 (worst). The pre-specified minimal clinically important difference is set at -1.5 point.
Symptoms of depression | 2 months
  Symptoms of depression will be assessed using the Hospital Anxiety and Depression questionnaire, depression subscore, before and after the rehabilitation program and after 1 year of the enrollement date. The score ranges from 0 (best) to 21 (worst). The pre-specified minimal clinically important difference is set at -1.5 point.
Symptoms of depression | One year
  Symptoms of depression will be assessed using the Hospital Anxiety and Depression questionnaire, depression subscore, before and after the rehabilitation program and after 1 year of the enrollement date. The score ranges from 0 (best) to 21 (worst). The pre-specified minimal clinically important difference is set at -1.5 point.
Cognitive function | 2 months
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA) test before, after the rehabilitation program and after 1 year of the enrollement date. Scores range from 0 to 30, with higher scores indicating better cognitive function. A score below 26 is considered indicative of mild cognitive impairement. The proportion of participants scoring below this threshold will be reported.
Cognitive function | One year
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA) test before, after the rehabilitation program and after 1 year of the enrollement date. Scores range from 0 to 30, with higher scores indicating better cognitive function. A score below 26 is considered indicative of mild cognitive impairement. The proportion of participants scoring below this threshold will be reported.
Objective physical activity | 2 months
  Objective physical activity will be measured using a triaxial accelerometer (Actigraph GTX3, Actigraph, Pensacola, FL, USA) worn by patients 10 days prior to study enrollement and 10 days after study completion. A measurement day will be considered valid if it includes at least 8 hours of use of the triaxial accelerometer. Physical activity assessment for a given patient will be considered valid if it includes at least 4 valid weekdays (i.e., more than 8 hours/day excluding weekends).
  The measurement will be adjusted for sunlight duration (included as a covariate in the analysis) Objective physical activity will also be measured one year after study enrollement.
Objective physical activity | One year
  Objective physical activity will be measured using a triaxial accelerometer (Actigraph GTX3, Actigraph, Pensacola, FL, USA) worn by patients 10 days prior to study enrollement and 10 days after study completion. A measurement day will be considered valid if it includes at least 8 hours of use of the triaxial accelerometer. Physical activity assessment for a given patient will be considered valid if it includes at least 4 valid weekdays (i.e., more than 8 hours/day excluding weekends).
  The measurement will be adjusted for sunlight duration (included as a covariate in the analysis) Objective physical activity will also be measured one year after study enrollement.
Sleep quality - Pittsburg sleep quality index | 2 months
  Sleep quality will be assessed using the Pittsburg Sleep Quality Index (PSQI) before and after the rehabilitation program and after 1 year of the enrollement date. Scores range from 0 to 21 with a lower score reflecting a better sleep quality.
Sleep quality - Pittsburg sleep quality index | One year
  Sleep quality will be assessed using the Pittsburg Sleep Quality Index (PSQI) before and after the rehabilitation program and after 1 year of the enrollement date. Scores range from 0 to 21 with a lower score reflecting a better sleep quality.
Sleep quality - Visual analog scale | 2 months
  Sleep quality will also be assessed using a Visual Analog Scale (VAS). Scores range from 0 to 10 with a higher score reflecting a better sleep quality.
Sleep quality - Visual analog scale | One year
  Sleep quality will also be assessed using a Visual Analog Scale (VAS). Scores range from 0 to 10 with a higher score reflecting a better sleep quality.
Auto-efficacy | 2 months
  Auto-efficacy will be measured using the french version of the self-efficacy for managing chronic disease scale before and after the rehabilitation program and after 1 year of the enrollement date. Possible score vary between 6 (weak self-efficacy) and 60 (high self-efficacy).
Auto-efficacy | One year
  Auto-efficacy will be measured using the french version of the self-efficacy for managing chronic disease scale before and after the rehabilitation program and after 1 year of the enrollement date. Possible score vary between 6 (weak self-efficacy) and 60 (high self-efficacy).
Autonomy support in health care settings | 2 months
  Autonomy support in health care settings will be assessed using the brief health care climate questionnaire (HCCQ). Possible scores vary from 6 (low autonomy support) to 42 (high autonomy support).
Autonomy support in health care settings | One year
  Autonomy support in health care settings will be assessed using the brief health care climate questionnaire (HCCQ). Possible scores vary from 6 (low autonomy support) to 42 (high autonomy support).
Adherence to exercise training | 2 months
  Adherence will be assessed as the ratio of completed sessions to prescribed sessions (24 sessions).
Adherence to self management | 2 months
  Adherence will be assessed as the ratio of completed sessions to prescribed sessions.
Environmental impact | 2 months
  The environmental impact will be assessed using the Climate Partner Hub software (Climate Partner®, Munich, Germany) and expressed as equivalent ton of carbon dioxide. The assessment will include a Life Cycle Assessment for each device used in both groups, data transmission and storage on cloud servers for home-based telerehabilitation, and transportation for both groups.
Exacerbations | One year
  Exacerbations will be collected during the rehabilitation program, after completion of the program and up to 1 year after enrollement date. They are categorized as follows:
  * Mild if they do not require any change in treatment or only an increase in bronchodilator use;
  * Moderate if they require the use of corticosteroids and/or antibiotics;
  * Severe if they result in hospitalization.
Hospitalization rate | One year
  Hospitalization rate will be collected during the rehabilitation program, after completion of the program and up to 1 year after enrollement date.
Death rate | One year
  Death rate will be collected during the rehabilitation program, after completion of the program and up to 1 year after enrollement date.
Health economic evaluation - Cost | 2 months
  A health economic evaluation will be conducted to assess the costs associated with each intervention.
Health economic evaluation - Cost | One year
  A health economic evaluation will be conducted to assess the costs associated with each intervention.
Health economic evaluation - Incremental cost utility ratio | 2 months
  A health economic evaluation will be conducted to assess the incremental cost utility ratio per quality-adjusted life year (QALY) gained
Health economic evaluation - Incremental cost utility ratio | One year
  A health economic evaluation will be conducted to assess the incremental cost utility ratio per quality-adjusted life year (QALY) gained
Health economic evaluation - Incremental cost effectiveness ratio | 2 months
  A health economic evaluation will be conducted to assess the incremental cost effectiveness ratio per endurance time gained
Health economic evaluation - Incremental cost effectiveness ratio | One year
  A health economic evaluation will be conducted to assess the incremental cost effectiveness ratio per endurance time gained

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Bonnevie, PhD, Principal Investigator — Association ADIR; Francis-Edouard Gravier, PhD, Study Chair — Association ADIR; Antoine Cuvelier, Prof, Study Chair — Association ADIR; Jean-François Muir, Prof, Study Chair — Association ADIR; Marc Beaumont, PhD, Study Chair — Centre Hospitalier des Pays de Morlaix; Guillaume Prieur, PhD, Study Chair — Groupe Hospitalier du Havre - Service de kinésithérapie; Yann Combret, PhD, Study Chair — Groupe Hospitalier du Havre - Service de kinésithérapie; Héloïse Baillet, PhD, Study Chair — Hôpital La Musse
Locations (4):
- France (4):
  - Groupe Hospitalier du Havre, Montivilliers
  - Centre Hospitalier des Pays de Morlaix, Morlaix
  - Association ADIR, Rouen
  - Hôpital La Musse, Saint-Sébastien-de-Morsent

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request for research purposes after publication. This includes de-identified data related to demographic characteristics, as well as endpoints published either in the main manuscript or any supplemental data. Requests should be sent to t.bonnevie@adir-hautenormandie.com
Time Frame: Data will be made available after publication.
Access Criteria: Data will be made available upon request, for research purpose. Request should be send to t.bonnevie@adir-hautenormandie.com

REFERENCES:
- [Background] McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD003793. doi: 10.1002/14651858.CD003793.pub3. PMID 25705944